CLINICAL TRIAL: NCT02514083
Title: A Pilot Phase II Study Using Ibrutinib and Short-Course Fludarabine in Previously Untreated Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: A Phase II Study Using Ibrutinib and Short-Course Fludarabine in Treatment-Naive CLL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150172; 15-H-0172 (Other: NIHCC)
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Bruton's tyrosine kinase inhibitor; Fludarabine; Immune modulation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ibrutinib and short-course fludarabine (Experimental): * Ibrutinib 420 mg PO daily for the duration of the study
  * Fludarabine 25 mg/m2/day IV on days 1-5 of cycles 3 and 4
  Interventions: Drug: Ibrutinib; Drug: Fludarabine

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib 420mg PO daily for the duration of the study.
  Other Names: Imbruvica
Drug: Fludarabine — Fludarabine 25 mg/m2/day IV on days 1-5 of cycles 3 and 4
  Other Names: Fludara

SUMMARY:
This is a pilot phase 2 study investigating the safety and efficacy of ibrutinib combined with short-course fludarabine in previously untreated CLL patients. Ibrutinib will be given daily until disease progression or intolerable side effects occur. Fludarabine will be given in cycles 3 and 4. The primary efficacy endpoint is the rate of complete response after 6 cycles or 24 weeks. The primary safety endpoint is the rate of treatment discontinuation after 6 cycles or 24 weeks.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) and/or small lymphocytic lymphoma (SLL) are tumors of B cells that often affect elderly patients. While the cause of CLL is still unclear, studies have indicated critical factors required for the tumor cells. First, CLL cells grow and survive because they receive signals through the B-cell receptor (BCR); and second, CLL cells benefit from interactions with other cells, especially T cells.

The stimulation through the BCR can be reduced with ibrutinib, which is an oral drug that selectively inhibits Bruton's tyrosine kinase (BTK). In clinical trials, ibrutinib demonstrated safety and high response rates in patients with high-risk disease. Ibrutinib has gained FDA approval as a treatment for CLL patients with 17p deletion and for those who had at least one prior therapy. However, single-agent ibrutinib has limitations; the drug does not eliminate all the tumor cells, and, with time, the tumor cells may become resistant. Therefore, a combination of ibrutinib with other drugs could be beneficial. Here we chose fludarabine because it is a well-tolerated drug that has been used widely to treat CLL. Also, fludarabine can kill both malignant B cells and T cells that support the growth of leukemia cells. With this approach, we hope to restore a healthier immune system.

This study will investigate the safety and efficacy of ibrutinib combined with fludarabine. This protocol is intended for previously untreated CLL patients. Ibrutinib will be given daily until disease progression or intolerable side effects occur. Fludarabine will be given only in cycles 3 and 4.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Men and women with histologically confirmed disease as defined by the following:

   * CLL: clonal B-lymphocytosis greater than or equal to 5,000 cells/microL .
   * SLL: lymphadenopathy with the tissue morphology of CLL but that are not leukemic, < 5,000 cells/microL.
   * Immunophenotypic profile or immunohistochemistry read by an expert pathologist as consistent with CLL. This will include CD5, CD19, and CD20 expression by the CLL cells typically also with CD23 expression, but CD23 negative cases may be included if there is an absence of t(11;14).
2. Active disease as defined by at least one of the following (IWCLL consensus criteria):

   * Weight loss greater than or equal to 10% within the previous 6 months
   * Extreme fatigue
   * Fevers of greater than 100.5 F for greater than or equal to 2 weeks without evidence of infection
   * Night sweats for more than one month without evidence of infection
   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia
   * Massive or progressive splenomegaly
   * Massive nodes or clusters or progressive lymphadenopathy
   * Progressive lymphocytosis with an increase of >50% over a 2-month period, or an anticipated doubling time of less than 6 months
3. Treatment naive CLL/SLL patients

   -Treatment-naive CLL indicates no prior anti-CLL therapy. Anti-CLL therapy includes chemotherapies, monoclonal antibodies, and targeted agents with known or reasonably expected anti-leukemic activity.
4. Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
5. Absolute neutrophil count (ANC) > 750/microL, platelets > 50,000/microL
6. Agreement to use acceptable methods of contraception during the study and for 90 days after the last dose of study drug if sexually active and able to bear or beget children. Female subjects of childbearing potential must have a negative serum pregnancy test upon study entry. Male and female subjects who agree to use both a highly effective method of birth control (eg, implants, injectables, combined oral contraceptives, some intrauterine devices, complete abstinence, or sterilized partner) and a barrier method (e.g. condoms, vaginal ring, sponge, etc.) during the period of therapy and for 90 days after the last dose of study drug.
7. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
8. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations)

EXCLUSION CRITERIA:

1. Transformed CLL, including Hodgkin and non-Hodgkin lymphoma
2. Active autoimmune hemolytic anemia or thrombocytopenia
3. Known bleeding disorders
4. Impaired hepatic function: Total bilirubin greater than or equal to 1.5 times upper limit of normal unless due to Gilbert's disease, aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than or equal to 2.5 times institutional upper limit of normal unless due to infiltration of liver, Child-Pugh class B or C
5. Impaired renal function: estimated glomerular filtration rate (GFR) < 30ml/min/1.73m(2) based on CKD-EPI
6. Life-threatening illness, medical condition or organ system dysfunction which, in the investigators opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib and fludarabine, or put the study outcomes at undue risk
7. Concomitant immunomodulatory therapy, chemotherapy, radiotherapy or experimental therapy
8. Active Hepatitis B or Hepatitis C infection
9. HIV infection
10. Female patients who are currently in pregnancy, or unwilling to use acceptable methods of contraception or refrain from pregnancy if of childbearing potential or currently breastfeeding. Male patients who are unwilling to follow the contraception requirements described in this protocol.
11. Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements.
12. Unable to understand the investigational nature of the study or give informed consent.
13. Individuals < 18 years old
14. Known hypersensitivity to any component of ibrutinib or fludarabine
15. Requires concomitant anticoagulation with Coumadin (warfarin) or other vitamin K antagonists.
16. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease-free for greater than or equal to 2 years or which will not limit survival to < 2 years
17. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
18. History of stroke or intracranial hemorrhage within 6 months before the first dose of study drug
19. Major surgery within 4 weeks of first dose of study drug
20. Currently active, clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, Class 3 or 4 congestive heart failure as defined by New York Heart Association Functional Classification, or a history of myocardial infarction or unstable angina, or acute coronary syndrome within 6 months of screening.
21. Subjects who received a strong cytochrome P450 (CYP) 3A inhibitor within 7 days prior to the first dose of ibrutinib or subjects who require continuous treatment with a strong CYP3A inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2034-10-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Itsara, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahn IE, Jerussi T, Farooqui M, Tian X, Wiestner A, Gea-Banacloche J. Atypical Pneumocystis jirovecii pneumonia in previously untreated patients with CLL on single-agent ibrutinib. Blood. 2016 Oct 13;128(15):1940-1943. doi: 10.1182/blood-2016-06-722991. Epub 2016 Aug 8. PMID 27503501
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-H-0172.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib With Fludarabine in Patients With CLL or SLL: Open-label study of ibrutinib and a short-course fludarabine in previously untreated participants with Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL). Ibrutinib is administered orally, 420 mg daily for duration of study. Fludarabine dose is 25 mg/m2/day on days 1-5 of cycles 3 and 4.
Period: Overall Study
Arm/Group | Ibrutinib With Fludarabine in Patients With CLL or SLL
Started | 29
Completed | 28
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib With Fludarabine in Patients With CLL or SLL
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Response at 24 Weeks
Description: Rate of complete response at 24 weeks or after 6 cycles. Response assessment was conducted according to the guidelines from the 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL).
Time Frame: 24 weeks
Population: Treatment-naive CLL or SLL patients
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib With Fludarabine in Patients With CLL or SLL
Number analyzed (Participants) | 28
Participants
  Complete response | 6
  Partial response with or without lymphocytosis | 21
  Stable disease | 1

2. Primary Outcome: Rate of Treatment Discontinuation Within the First 24 Weeks
Description: Rate of treatment discontinuation within the first 24 weeks or 6 cycles due to intolerable side effects from study therapy
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib With Fludarabine in Patients With CLL or SLL
Number analyzed (Participants) | 29
Participants
  Treatment discontinued within 24 weeks | 1
  Treatment continued for 24+ weeks | 28

ADVERSE EVENTS:
Time Frame: From treatment initiation until the last follow-up on study or death, whichever occurred first, assessed up to 4 years
Description: The AE reporting period for this study begins when the participant takes the first dose of study drug and continues until the last follow-up on the study. Participants will continue on study until disease progression or intolerable side effects occur.
Groups:
- Ibrutinib With Fludarabine in Patients With CLL or SLL: Open-label study of ibrutinib and a short-course fludarabine in previously untreated participants with Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL). Ibrutinib is administered orally, 420 mg daily for days 1-28 from Cycle 1 up to Cycle 27. Fludarabine dose is 25 mg/m2/day on days 1-5 of cycles 3 and 4.
Arm/Group | Ibrutinib With Fludarabine in Patients With CLL or SLL
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 14/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib With Fludarabine in Patients With CLL or SLL (N=29)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Post-operative Hemorrhage (Epistaxis) (Injury, poisoning and procedural complications) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vulvar intraepithelial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Triple negative Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib With Fludarabine in Patients With CLL or SLL (N=29)
White blood cell decreased (Investigations) | 19 (19)
Leukocytosis (Blood and lymphatic system disorders) | 14 (14)
Platelet count decresaed (Investigations) | 14 (14)
Neutrophil count decresaed (Investigations) | 12 (12)
Bruising (Injury, poisoning and procedural complications) | 19 (19)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (12)
Fatigue (General disorders) | 9 (9)
Hypertension (Vascular disorders) | 9 (9)
Pain (General disorders) | 7 (7)
Peripheral edema (General disorders) | 7 (7)
Brittle nails (Skin and subcutaneous tissue disorders) | 8 (8)
Petechiae (Skin and subcutaneous tissue disorders) | 6 (6)
Shingles (Infections and infestations) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 5 (5)
Headache (Nervous system disorders) | 4 (4)
Alanine or aspartate aminotransferase increased (Investigations) | 4 (4)
Lung infection (Infections and infestations) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 14 (14)
Lymphocyte count increased (Investigations) | 8 (8)
Nausea (Gastrointestinal disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Creatinine increased (Investigations) | 4 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Flu like symptoms (General disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Hematoma (Blood and lymphatic system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Infections and infestations: other (Infections and infestations) | 2 (2)
Productive cough (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Weight gain (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT02514083/Prot_SAP_000.pdf